CLINICAL TRIAL: NCT06210906
Title: Gastric Volume Following Sips of Water Intake Within 1 Hour in Preoperative Fasting Elderly Patients; Observational Study
Brief Title: Gastric Volume Following Sips of Water Intake
Status: Not yet recruiting | Type: Observational
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Professor, SMG-SNU Boramae Medical Center
Other Study IDs: 2024-1
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Stomach Filling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sips of water: Patients taking sips of water within 1 hour in preoperative fasting
  Interventions: Other: Assessment of gastric volume
- No sips of water: Patients not taking sips of water within 1 hour in preoperative fasting
  Interventions: Other: Assessment of gastric volume

INTERVENTIONS:
Other: Assessment of gastric volume — Gastric volume is assessed using ultrasound.

SUMMARY:
We aim to observe whether drinking of sips of water within 1 hour before surgery significantly affects the gastric volume.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years old undergoing elective surgery under general anesthesia

Exclusion Criteria:

* History of gastric surgery
* Anatomical anomaly, diseases, or mass in the stomach

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 65 years old undergoing elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-26 (Estimated); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Gastric volume | Immediately before induction of anesthesia
  Gastric volume is assessed using ultrasound in the supine and right lateral decubitus position.